CLINICAL TRIAL: NCT02473003
Title: Physical Training and Cancer- Effects and Understanding of Mechanisms for Prevent and Minimizing Cancer Related Fatigue, Improve Quality of Life and Disease Outcome
Brief Title: Physical Training and Cancer-a Multicenter Clinical Trial
Acronym: Phys-Can
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Cancer Society (Other); Nordic Cancer Union (Other); Linkoeping University (Other Government); Lund University (Other); University of Agder (Other); Copenhagen University Hospital, Denmark (Other); Norwegian School of Sport Sciences (Other); Amsterdam UMC, location VUmc (Other); University of Amsterdam (Other); University of Leeds (Other)
Responsible Party: Principal Investigator, Karin Nordin, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0273401, CAN2012/631,621
Record Dates: First submitted 2014-10-10; First posted 2015-06-16 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Colorectal Cancer; Prostate Cancer
Keywords: Breast cancer; prostate cancer; colorectal cancer; fatigue; physical exercise; randomised trial; intervention
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Fatigue; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- High intensity (Experimental): high intensity exercise 80-90%
  Interventions: Behavioral: high intensity exercise
- Low/Medium intensity (Experimental): low/medium intensity exercise 40-50%
  Interventions: Behavioral: low/medium intensity exercise
- High Intensity with BM (Experimental): high intensity exercise with Behavioral medicine strategies¨ 80-90%
  Interventions: Behavioral: high intensity exercise; Behavioral: Behavioral medicine strategies
- Low/Medium intensity with BM (Experimental): low/medium intensity exercise with Behavioral medicine strategies 40-50%
  Interventions: Behavioral: low/medium intensity exercise; Behavioral: Behavioral medicine strategies

INTERVENTIONS:
Behavioral: high intensity exercise — high intensity exercise 80-90%
  Arms: High Intensity with BM; High intensity
Behavioral: low/medium intensity exercise — low/medium intensity exercise 40-50%
  Arms: Low/Medium intensity; Low/Medium intensity with BM
Behavioral: Behavioral medicine strategies — Motivational and self-regulatory behavioral medicine support strategies
  Arms: High Intensity with BM; Low/Medium intensity with BM

SUMMARY:
Excessive tiredness (fatigue) is a common problem in cancer patients and can affect quality of life negatively. There is limited knowledge about the physical mechanisms that cause fatigue, and there is no medical treatment. Physical activity can reduce the inconvenience, but the investigators need to learn more about the type and intensity of exercise that works the best as well as how to motivate patients to exercise. The overall aim, is to evaluate the efficacy and cost-effectiveness of individually tailored high (H) and low/medium (LM) intensity physical training, with or without behavioural medicine (BM) support strategies, during adjuvant oncological treatment on; Cancer Related Fatigue (CRF),Quality of Life (QoL), mood disturbance, adherence to the cancer treatment, adverse effects, disease outcome, return to a daily life after completed treatment and return to work. The investigators will also describe changes in inflammatory markers and cytokines related to physical training and gene expressions following training to investigate whether these serve as mediators for the effects of physical training on CRF and QoL. This will be evaluated in newly diagnosed breast, colorectal and prostate cancer patients during adjuvant therapy at three different centres in Sweden; Uppsala, Lund/Malmö and Linköping. A 2x2 factorial design will be used, 600 patients will be randomised to H, H+BM, LM or LM+BM. Patients will train two times per week during 6 months. This project will give; new knowledge about aspects for individuals to gain improved well-being and quality of life, facilitated return to work, and possibly reduced risk of cancer recurrence. This in turn would result in lower burden on the health care system, reduced societal costs and have a positive impact on public health. Implementation of the results into clinical practice will be facilitated by the close collaboration between researchers and clinicians, and the fact that the study is performed in clinical settings.

DETAILED DESCRIPTION:
Purpose and Aims The main aim is to determine the effects of high or low intensity physical training with or without integrated behavioral medicine support strategies to prevent and minimize cancer related fatigue (CRF), improve health related quality of life (QoL) and to understand the role of inflammation and cytokines in the development and maintenance of CRF, as well as to increase knowledge with respect to cost-effectiveness of rehabilitation programs. This will be evaluated in newly diagnosed breast, colorectal and prostate cancer patients during adjuvant therapy at three different centers in Sweden; Uppsala, Lund/Malmö and Linköping and one in Norway.

More specifically, the investigators' objectives are to:

1. Investigate the effects of high intensity training compared to low intensity training on patient reported outcomes (CRF as primary endpoint), chemotherapy/radiation completion rates, medical (oncology) adverse effects, physical activity and daily function, during adjuvant treatment and at long-term-follow up. In addition, effects on the course of disease (e.g time to relapse).
2. Investigate if supplemental behavioural medicine support strategies increase adherence to exercise during adjuvant therapy and further if they increase the maintenance of physical activity behaviours and decrease sedentary time in the long run.
3. Explore the role of changes in inflammatory markers and cytokines related to physical training and following training to investigate whether these serve as mediators for the effects of physical training on CRF and QoL.
4. Pursue the investigation of a direct role of cytokines secreted from the working muscles, in inhibiting cancer cell growth and inducing apoptosis.
5. Evaluate health economic issues; cost effectiveness of the interventions, health production and individual wellbeing.

In Phys-Can, the investigators will implement rigorously designed and adequately powered randomized longitudinal multicenter clinical trials, with physical training and behavioral medicine support interventions. The highly multi- and interdisciplinary and international consortium behind this proposal is in an excellent position to perform international and interdisciplinary competence- and network-building activities to generate valid, high quality data covering all areas included in the project, from basic biomedical data to patient reported outcomes (PROs), i.e. from bench to bedside. This is unique in health care sciences.

Study design A 2x2 factorial design will be used. With this design the investigators can study main effects and interactions between factors (groups). Patients will be randomized to one of the following groups; A) individually tailored high intensity training twice a week with (H+BM) or without behavioral medicine support strategies (H) or B) individually tailored low intensity training twice a week with (L+BM) or without behavioral medicine support strategies (L).

Study sample/procedure Patients, who are recently diagnosed with breast cancer, colorectal cancer or prostate cancer and scheduled for adjuvant therapy at Uppsala, Lund/Malmö, Linköping and Haukeland University hospitals will be consecutively included in the study. Based on the power calculation, 612 patients will be included.

All patients will exercise twice a week during 6 months which is equal to the most extensive adjuvant treatment period. It is also an optimal period to achieve physical training effects and to establish physical activity behavior. Physical training under the guidance of trained coaches will be offered twice a week. Training intensity is 40-50% (low intensity group) or 80-90% (high intensity group) of maximal cardiorespiratory fitness/muscular strength. Physical training sessions consist of both cardiorespiratory and resistance exercise. Every four week, progress from resistance training is evaluated by means of a strength test, and absolute intensity is adjusted accordingly Motivational and self-regulatory behavioral medicine support strategies (motivational and self-regulatory strategies) will be provided for the H+BM and the L+BM groups i.e. strategies to enhance engagement in the high and low intensity exercise programs respectively, and to maintain health enhancing physical activity after the completion of the programs.

ELIGIBILITY:
Inclusion Criteria:

* understand and talk Swedish.
* patients with breast cancer who receive neoadjuvant / adjuvant chemotherapy and / or adjuvant radiotherapy and / or adjuvant endocrine treatment.
* patients with colorectal cancer who receive adjuvant chemotherapy.
* patients with prostate cancer who receive neoadjuvant / adjuvant endocrine treatment with the addition of curative radiation therapy.

Exclusion Criteria:

* Patients unable to perform basic activities of daily living.
* Patients with cognitive disorders such as dementia and severe psychiatric illness.
* Patients with disabilities that may prevent physical activity: (eg, unstable angina, heart failure, chronic obstructive pulmonary disease, orthopedic and neurological diseases).
* Breast cancer stage IIIb.
* Undergoing treatment for other types of malignant disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-03; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue | post oncol treatment (expected time frame 6-8 weeks), 6 month, 1,2,5 years
  Multi Dimensional Fatigue Inventory (MFI),

SECONDARY OUTCOMES:
Change in Quality of Life | post oncol treatment (expected time frame 6-8 weeks), 6 month, 1,2,5 years
  The European Organisation for Research and Treatment of Cancer (EORTC)EORTC-QLQ30
Change in Mood disturbance | post oncol treatment (expected time frame 6-8 weeks), 6 month, 1,2,5 years
  Hospital Anxiety and Depression Scale- (HADs)
Change in Function in Daily life | 6 months,1, 2, 5 years
  WHO Disability Assessment Schedule
Change in pain | post oncol treatment (expected time frame 6-8 weeks), 6 month, 1,2,5 years
  Brief Pain Inventory
Change in Cardio respiratory fitness | 6 month
  maximal oxygen uptake (VO2 max test)
Change in Muscle strength | 6 months
  One Repetition Maximum Lower extremities: One Repetition Maximum (leg press)
Health Economy | 12 months
  Euroqol- (EQ5D)
Cancer recurrence | 10 year
  number of patients with recurrence
Sleep | 6 months
  Insomnia severe index
Health Economy register | 12 months
  register data
Cancer recurrence | 6 months, 1, 2, 5, 10 years
  Medical records
Treatment completion rate | 1, 2, 5, 10 year
  Medical records

CONTACTS AND LOCATIONS:
Overall Officials: Karin Nordin, Professor, Principal Investigator — Uppsala University

REFERENCES:
- [Derived] Mazzoni AS, Helgesen Bjorke AC, Stenling A, Borjeson S, Sjovall K, Berntsen S, Demmelmaier I, Nordin K. The Role of Long-Term Physical Activity in Relation to Cancer-Related Health Outcomes: A 12-Month Follow-up of the Phys-Can RCT. Integr Cancer Ther. 2023 Jan-Dec;22:15347354231178869. doi: 10.1177/15347354231178869. PMID 37358262
- [Derived] Mazzoni AS, Strandberg E, Borjeson S, Sjovall K, Berntsen S, Demmelmaier I, Nordin K. Reallocating sedentary time to physical activity: effects on fatigue and quality of life in patients with breast cancer in the Phys-Can project. Support Care Cancer. 2023 Feb 4;31(2):151. doi: 10.1007/s00520-023-07614-9. PMID 36738358
- [Derived] Henriksson A, Strandberg E, Stenling A, Mazzoni AS, Sjovall K, Borjeson S, Raastad T, Demmelmaier I, Berntsen S, Nordin K. Does inflammation markers or treatment type moderate exercise intensity effects on changes in muscle strength in cancer survivors participating in a 6-month combined resistance- and endurance exercise program? Results from the Phys-Can trial. BMC Sports Sci Med Rehabil. 2023 Jan 19;15(1):8. doi: 10.1186/s13102-023-00617-3. PMID 36658635
- [Derived] Schauer T, Henriksson A, Strandberg E, Lindman H, Berntsen S, Demmelmaier I, Raastad T, Nordin K, Christensen JF. Pre-treatment levels of inflammatory markers and chemotherapy completion rates in patients with early-stage breast cancer. Int J Clin Oncol. 2023 Jan;28(1):89-98. doi: 10.1007/s10147-022-02255-0. Epub 2022 Oct 21. PMID 36269530
- [Derived] Brooke HL, Mazzoni AS, Buffart LM, Berntsen S, Nordin K, Demmelmaier I. Patterns and determinants of adherence to resistance and endurance training during cancer treatment in the Phys-Can RCT. BMC Sports Sci Med Rehabil. 2022 Aug 13;14(1):155. doi: 10.1186/s13102-022-00548-5. PMID 35964124
- [Derived] Mazzoni AS, Brooke HL, Berntsen S, Nordin K, Demmelmaier I. Effect of self-regulatory behaviour change techniques and predictors of physical activity maintenance in cancer survivors: a 12-month follow-up of the Phys-Can RCT. BMC Cancer. 2021 Nov 25;21(1):1272. doi: 10.1186/s12885-021-08996-x. PMID 34823494
- [Derived] Schauer T, Mazzoni AS, Henriksson A, Demmelmaier I, Berntsen S, Raastad T, Nordin K, Pedersen BK, Christensen JF. Exercise intensity and markers of inflammation during and after (neo-) adjuvant cancer treatment. Endocr Relat Cancer. 2021 Mar;28(3):191-201. doi: 10.1530/ERC-20-0507. PMID 33608485
- [Derived] Mazzoni AS, Brooke HL, Berntsen S, Nordin K, Demmelmaier I. Exercise Adherence and Effect of Self-Regulatory Behavior Change Techniques in Patients Undergoing Curative Cancer Treatment: Secondary Analysis from the Phys-Can Randomized Controlled Trial. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420946834. doi: 10.1177/1534735420946834. PMID 32909467
- [Derived] Johnsson A, Demmelmaier I, Sjovall K, Wagner P, Olsson H, Tornberg AB. A single exercise session improves side-effects of chemotherapy in women with breast cancer: an observational study. BMC Cancer. 2019 Nov 8;19(1):1073. doi: 10.1186/s12885-019-6310-0. PMID 31703567
- [Derived] Berntsen S, Aaronson NK, Buffart L, Borjeson S, Demmelmaier I, Hellbom M, Hojman P, Igelstrom H, Johansson B, Pingel R, Raastad T, Velikova G, Asenlof P, Nordin K. Design of a randomized controlled trial of physical training and cancer (Phys-Can) - the impact of exercise intensity on cancer related fatigue, quality of life and disease outcome. BMC Cancer. 2017 Mar 27;17(1):218. doi: 10.1186/s12885-017-3197-5. PMID 28347291